CLINICAL TRIAL: NCT06625853
Title: Supplementary Use of the XP-Endo Finisher on Postoperative Pain in Retreatment Cases Using Mtwo R Files (Randomized Clinical Trial)
Brief Title: XP-Endo Finisher on Postoperative Pain in Retreatment Cases Using Mtwo R Files
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0738-08/2023
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Dental Pain; Endodontically Treated Teeth
MeSH Terms: conditions — Toothache; Tooth, Nonvital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mtwo R files without Xp-endo finisher file. (Experimental)
  Interventions: Other: Mtwo R files
- Mtwo R files followed by Xp-Endo finisher file (Experimental)
  Interventions: Other: Mtwo R files with Xp-Endo finisher file

INTERVENTIONS:
Other: Mtwo R files with Xp-Endo finisher file — XP-endo Finisher file will be inserted without rotation into the root canals filled with 2.5% NaOCl and will be activated (800 rpm; torque of 1 N.cm) for
  1 min in each canal using slow and gentle 7-8 mm lengthwise movements.
  Arms: Mtwo R files followed by Xp-Endo finisher file
Other: Mtwo R files — obturation material will be removed using Mtwo R (VDW, Munich, Germany)files attached to an endodontic motor (Ecube, seachin, Korea) with a constant speed of 280 rpm, as suggested by the manufacturer. Mtwo R 25/0.05 will be used to empty the coronal and middle thirds of the root. Mtwo R 15/0.05 will be used to reach the working length.
  Arms: Mtwo R files without Xp-endo finisher file.

SUMMARY:
Introduction: Postoperative pain is one of the most critical issues in our daily practice. , postoperative pain control is essential for patient satisfaction and comfort. When primary root canal treatment fails, root canal retreatment aims to heal apical periodontitis.

Aim of study: To compare between postoperative pain (POS) after endodontic retreatment using NI-TI rotary files Mtwo R alone and in conjunction with XP endo finisher .

Materials and Methods: This research is a randomized clinical trial conducted in a parallel design on 50 patients needing retreatment. They will be divided into two groups, group 1 retreatment with Mtwo R, group 2 retreatment with Mtwo R followed by Xp - Endo finisher. Postoperative pain levels will be evaluated at 24 hours, 48 hours, 72 hours, and 7 days following the removal of the obturation mat erial. The assessment of pain will be done through clinical examination, The Defense and veterans pain rating scale (DVPRS) and by the intake of pain killer

ELIGIBILITY:
Inclusion Criteria:

* Teeth with mature apices.
* Patients with no systemic diseases.
* No analgesic, anti-inflammatory, or antibiotic intake during 7 days before treatment.
* Teeth showing failure of initial root canal treatment and radiograph evidence of periapical bone destruction

Exclusion Criteria:

* Multi rooted teeth.
* Teeth with open apices.
* Teeth with cracks, calcification, root caries, fractures, external or internal resorption.
* Allergies to local anesthetic agents.
* Presence of severe pain and/or acute apical abscesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Change in pain | 24-hours,48-hours,72hours and 7 days
  Word descriptors are attached to each number on the DVPRS
  0 = No pain
  1. = Hardly noticeable pain
  2. = Noticeable pain, but does not interfere with activities
  3. = Somewhat distracting pain
  4. = Distracting pain, but does not affect normal activities
  5. = Pain interrupts some activities
  6. = Hard to ignore pain, avoidance of daily activities
  7. = Pain is the main focus of attention, prevents daily activities
  8. = Awful pain, difficult to do anything
  9. = Unbearable pain, cannot do anything
  10. = As bad as pain can be, nothing else matters

SECONDARY OUTCOMES:
change in analgesics intake according to severity of pain according to WHO Analgesic Ladder | 24-hours,48-hours,72hours and 7 days
  First Step - Mild pain: non-opioid analgesics such as nonsteroidal antiinflammatory drugs (NSAIDs) or acetaminophen with or without adjuvants.
  * Second Step - Moderate pain: weak opioids (hydrocodone, codeine, tramadol) with or without non-opioid analgesics and with or without adjuvants.
  * Third Step - Severe and persistent pain: potent opioids (morphine, methadone, fentanyl, oxycodone, buprenorphine, tapentadol, hydromorphone, oxymorphone) with or without non-opioid analgesics, and with or without adjuvants.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt